CLINICAL TRIAL: NCT04559802
Title: Submerged Versus Non-Submerged Healing of Implants Subjected to Contour Augmentation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Theofilos Koutouzis, Principal Investigator, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-341
Record Dates: First submitted 2020-09-06; First posted 2020-09-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transmucosal (Non-Submerged) (Experimental): Flaps will be adapted to the healing abutments for a trans-mucosal healing up on closure
  Interventions: Procedure: Transmucosal Technique
- Submerged (Active Comparator): Flaps will be advanced to achieve primary wound closure.
  Interventions: Procedure: Submerged Technique

INTERVENTIONS:
Procedure: Transmucosal Technique — Dental implant will be placed in transmucosal manner (Healing abutment is exposed in the mouth).
  Other Names: Non-submerged technique
  Arms: Transmucosal (Non-Submerged)
Procedure: Submerged Technique — Dental implant will be installed in submerged manner (implant is completed covered by soft tissue).
  Arms: Submerged

SUMMARY:
It is a randomized controlled trial to evaluate two surgical techniques for dental implant placement simultaneously with bone augmentation.

DETAILED DESCRIPTION:
Implants receiving Contour Augmentations at the time of placement are randomized into two groups, submerged and non submerged. Healing is evaluated at 4 months post op compared to the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 21 years - ASA I or II.
* Patient's willingness to participate in this study.
* Availability for 4-month follow-up.
* Absence of active periodontal disease.
* Single tooth replacement is needed with simultaneous contour augmentation.
* Available pre-operative CBCT study.
* Extraction of tooth at least 8 weeks prior to planned implant therapy.

Exclusion Criteria:

* Pregnancy at the screening visit.
* Smoking more than 10 cig/day.
* Active infection at the site of surgery (teeth involved).
* Multiple missing teeth adjacent to each other (long span edentulous area).
* Vertical bone defect less than 2mm (intra surgical assessment)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Hard tissue healing around dental implants | 4 months
  bone healing around Submerged and Non-submerged dental implants will be measured by Periodontal probe and radiographs. A Mann-Whitney U Test will be used to calculate bone healing changes. To evaluate bone healing Mean values, standard deviations and frequencies will be calculated.

SECONDARY OUTCOMES:
Soft tissue healing around dental implants | 4 months
  Soft tissue healing around Submerged and Non-submerged dental implants. Fisher's exact test will be used to evaluate soft tissue healing changes through analyzing the measurements obtained by periodontal probe and radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Sofos, DDS, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova South Eastern university, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No